CLINICAL TRIAL: NCT06351306
Title: A Phase II Open-Label, Single Center Trial of Oral Decitabine-Cedazuridine (DEC-C) (Inqovi®) in Combination With Thioguanine (Tabloid®) in Patients With Relapsed or Refractory (R/R) Acute Myeloid Leukemia (AML)
Brief Title: DEC-C and Thioguanine for R/R AML
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficultly enrolling
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAU5915
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: Myeloid Neoplasm; Cancer
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasms | interventions — Thioguanine; decitabine and cedazuridine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Safety Lead-In (Experimental): Groups of participants will receive different doses of thioguanine and decitabine-cedazuridine to identify the highest doses that can be given safely. The highest doses that are safe will then be used in the phase II portion of the clinical trial. If no dose is found to be safe, the study will be stopped.
  A phase II expansion cohort will be enrolled to further explore the combination's anti-leukemia activity and safety and will proceed at the maximum tolerated dose defined in the initial Safety Cohort.
  Interventions: Drug: Thioguanine (Tabloid ®); Drug: DecitabineCedazuridine (Inqovi ®)

INTERVENTIONS:
Drug: Thioguanine (Tabloid ®) — 60-80mg/m^2 oral tablet
Drug: DecitabineCedazuridine (Inqovi ®) — 35 mg decitabine and 100 mg cedazuridine oral tablet

SUMMARY:
The purpose of this study is to find out if oral decitabine-cedazuridine (Inqovi®) is effective, safe, and able to be tolerated without severe side effects when given with thioguanine (Tabloid®) in patients with acute myeloid leukemia (AML) whose disease has returned or did not respond to treatment (relapsed or refractory).

This is a "phase II trial with a safety lead-in." The goal of the lead-in portion of the study is to make sure participants are getting the highest dose of medications that are safe. If too many serious side effects are seen with the dose previously studied, some additional patients may be treated with a lower dose to make sure that this dose is safe.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is a cancer of the blood and bone marrow with a 5-year survival rate of 47.5% for patients less than age 65 years and only an 8.2% survival for those 65 and older, based on data from the Surveillance, Epidemiology, and End Results (SEER) program of the National Cancer Institute. Despite some advances in treatment, most patients will relapse, and treatment remains limited, especially for patients that progress on the standard of care. The expected response rate to salvage chemotherapy is only 10-20% with a median survival typically of less than 6 months. The need for new, effective, and well-tolerated treatments is clear.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years of age
2. Patients must have histologically and cytologically confirmed R/R AML according to the World Health Organization classification based on documented bone marrow biopsy or peripheral blood specimens, with the exception of acute promyelocytic leukemia

   1. Relapsed AML is defined as the detection of ≥5% blasts in the bone marrow or reappearance of leukemic blasts in the peripheral blood in a patient with prior remission
   2. Refractory AML is defined as the failure to obtain a CR, CRh, or CRi after at least two courses of intensive induction (including hypomethylating agent plus venetoclax induction) or at least six cycles of a hypomethylating agent-based regimen (except venetoclax combinations as above)
3. Able to provide informed consent
4. Eastern Cooperative Oncology Group (ECOG) performance score of 0 to 2 or Karnofsky ≥60%
5. Adequate organ function defined by the following parameters:

   1. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤5x the upper limit of normal (ULN)
   2. Bilirubin ≤2x the ULN unless due to known Gilbert's disease or hemolysis due to blood transfusion
   3. Calculated glomerular filtration rate (GFR) of ≥ 30 mL/min/1.73 m2
6. Prior hypomethylating agent is allowed
7. Female patients of childbearing potential must not be nursing or planning to become pregnant and require a negative urine or serum pregnancy test within 30 days of study therapy.
8. Female patients of childbearing potential must be willing to use at least 1 method of highly effective contraception during the study. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
9. Male patients treated or enrolled who are sexually active must agree to adequate contraception use and refrain from sperm donation throughout the duration of the study, and up to 4 months after completion of thioguanine and decitabine-cedazuridine.
10. Willing to provide pretreatment bone marrow aspirate and biopsies samples as well as subsequent bone marrow aspirate and biopsies samples during the study.
11. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Previously received thioguanine
2. Any anti-leukemic therapy, including investigational therapies, within 14 days of study treatment initiation. Hydroxyurea for blood count control is allowed throughout induction cycle(s)
3. Prior allogeneic hematopoietic stem cell transplantation within 3 months of study enrollment; active graft versus host disease
4. Clinical suspicion for active central nervous system (CNS) involvement by AML; previously treated CNS involvement is allowed
5. Second malignancy requiring treatment within 6 months of study enrollment, with the exception of non-melanoma skin cancers or cancers requiring hormonal therapy only
6. Active, uncontrolled infection
7. Human immunodeficiency virus (HIV) not controlled by standard therapy
8. Active hepatitis B or C infection. Participants whose infections are controlled with antiviral therapy are allowed.
9. Significant medical diseases or comorbidities, in the opinion of the investigator, that would preclude the safe participation in the study
10. Known hypersensitivity to DEC-C or thioguanine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Composite Complete Remission (CRc) Rate | Up to 3 years
  This rate will be calculated from rate of complete remission (CR) plus CR with partial hematologic recovery (CRh) plus CR with incomplete hematologic recovery (CRi), according to the European LeukemiaNet (ELN) 2022 criteria.

SECONDARY OUTCOMES:
Duration of Remission | Up to 3 years
  This is defined as the time from CRc until relapse or death from any cause, whichever is first.
Time to Complete Remission (CR) | Up to 3 years
  This is defined as time from therapy initiation until CRc.
Overall Survival (OS) | Up to 3 years
  This is defined as the duration of time from randomization to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph G. Jurcic, MD, Principal Investigator — Columbia University